CLINICAL TRIAL: NCT03102632
Title: A Clinical Trial of Water Therapy for Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1701017921
Record Dates: First submitted 2017-03-27; First posted 2017-04-06 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Autosomal Dominant Polycystic Kidney
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Intervention Model Description: Participants will have a period of usual fluid intake and a period of increased water intake over the course of the study.
Who Masked: Outcomes Assessor
Masking Description: The radiologist measuring kidney volumes will be masked to the study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Water Intake (No Intervention): For the first 6 months of the study, the participants will continue their usual water intake.
- High Water Intake (Experimental): After a 6 month period of usual water intake, a high water intake daily amount will be prescribed for 1 year.
  Interventions: Other: High Water Intake

INTERVENTIONS:
Other: High Water Intake — After 6 months of usual, unchanged diet and fluid intake, participants will be asked to increase the daily fluid intake based on the principal investigator's prescription. The actual amount of extra water prescribed will depend on the results of the participant's 24 hour urine test.
  Arms: High Water Intake

SUMMARY:
Patients affected by Autosomal Dominant Polycystic Kidney Disease (ADPKD) need a safe and effective long-term treatment regimen. Unfortunately, there are still no disease-specific treatment for ADPKD approved in the US. A rational step towards identifying such agents is to test therapies that have a proven safety profile with mechanisms of action that can counter the disease progression.

The purpose of this study is to investigate whether drinking increased amounts of water (water loading) might slow down polycystic kidney growth or kidney function decline. Water loading can cause the suppression of a pathway that causes fluid buildup and cyst growth. High water intake has been safely used in the clinical setting, such as in the case of kidney stone therapy. New York State tap water is widely available and safe, making it highly cost-effective as well.

DETAILED DESCRIPTION:
The study will involve 11 visits to the study site over 19 months. Participants will need to follow specific dietary and fluid recommendations. There will be physical examinations and medical history assessments at each visit. Testing will include undergoing magnetic resonance imaging (MRI), blood and urine tests. Study participants will be compensated for their time. Detailed study procedures will be reviewed upon contact with the study team.

ELIGIBILITY:
Inclusion Criteria:

* pre-existing diagnosis of Autosomal Dominant Polycystic Kidney Disease
* estimated glomerular filtration rate of 40 ml/min or greater
* urine osmolality > 400 mOsm/L

Exclusion Criteria:

* estimated glomerular filtration rate less than 40 ml/min
* low blood sodium levels
* syndrome of inappropriate diuretic hormone
* use of thiazide diuretics or selective serotonin reuptake inhibitors (SSRIs)
* use of tolvaptan, another vasopressin receptor antagonist, vasopressin agonists or dDAVP
* contraindications to magnetic resonance imaging (MRI) (pacemakers, defibrillators, implanted electronic devices, metallic foreign body)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in total kidney volume, as measured from magnetic resonance imaging | 18 months
  Total kidney volumes will be measured before and after the period of high water intake. Kidney volume growth with high water intake will be compared to baseline kidney volume growth.

SECONDARY OUTCOMES:
Kidney function change | 18 months
  Blood creatinine levels will be measured and compared before and after the high water intake period.
Change in urine and blood markers of response to high water intake | 18 months.
  Blood and urine biomarkers of response to high water intake will be measured before and after the period of high water intake.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Prince, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dev H, Zhu C, Barash I, Blumenfeld JD, He X, RoyChoudhury A, Wu A, Prince MR. Feasibility of Water Therapy for Slowing Autosomal Dominant Polycystic Kidney Disease Progression. Kidney360. 2024 May 1;5(5):698-706. doi: 10.34067/KID.0000000000000428. Epub 2024 Apr 1. PMID 38556640